CLINICAL TRIAL: NCT01513590
Title: A 26-week, Randomised, Open-label, Multinational, Treat-to-target Trial Comparing Efficacy and Safety of Insulin Degludec/Insulin Aspart (IDegAsp) Twice Daily (BID) and BIAsp 30 BID Both With Metformin in Insulin naïve Subjects With Type 2 Diabetes Mellitus Inadequately Controlled on Metformin Monotherapy or Metformin in Combination With One Additional Oral Antidiabetic Drug (OAD)
Brief Title: A Trial Comparing Efficacy and Safety of Insulin Degludec/Insulin Aspart and BIAsp 30 in Insulin naïve Subjects With Type 2 Diabetes
Acronym: BOOST™
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN5401-3940; 2011-001712-61 (EudraCT Number); U1111-1120-5633 (Other: WHO)
Record Dates: First submitted 2012-01-16; First posted 2012-01-20 (Estimated); Results first posted 2015-11-20 (Estimated); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin degludec, insulin aspart drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IDegAsp BID (Experimental)
  Interventions: Drug: insulin degludec/insulin aspart
- BIAsp 30 BID (Active Comparator)
  Interventions: Drug: insulin degludec/insulin aspart

INTERVENTIONS:
Drug: insulin degludec/insulin aspart — Administered s.c. (under the skin) twice daily. Dose individually adjusted. Pre-trial metformin treatment to be continued.

SUMMARY:
This trial is conducted in Africa, Asia and Europe. The aim of the trial is to compare the efficacy and safety of insulin degludec/insulin aspart and BIAsp 30 (biphasic insulin aspart 30) in insulin naïve subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities. (Trial-related activities are any procedure that would not have been performed during normal management of the subject)
* Type 2 diabetes mellitus (diagnosed clinically) for at least 24 weeks prior to screening
* Current treatment: metformin monotherapy or metformin in any combination with one of the following oral anti-diabetic drugs (OADs): insulin secretagogue (sulfonylurea or glinide), dipeptidyl peptidase IV (DPP-IV) inhibitor, alpha-glucosidase inhibitors for at least 12 weeks prior to randomisation (Visit 2) with the minimum doses stated: - Metformin: alone or in combination (including fixed combination) 1500 mg daily, or maximum tolerated dose (at least 1000 mg daily), - Insulin secretagogue (sulphonylurea or glinide): minimum half of the daily maximum dose according to local labelling, - DPP-IV inhibitor: minimum 100 mg daily or according to local labelling, - Alpha-glucosidase-inhibitors: minimum half of the daily maximum dose or maximum tolerated dose
* Insulin naïve subject; allowed is: Previous short term insulin treatment up to 14 days
* Insulin naïve subject; allowed is: Treatment during hospitalization or during gestational diabetes is allowed for periods longer than 14 days)
* HbA1c (glycosylated haemoglobin) between 7.0-10.0 % (both inclusive) by central laboratory analysis
* Body mass index (BMI) below or equal to 40.0 kg/m^2

Exclusion Criteria:

* Treatment with thiazolidinediones (TZDs) or glucagon like peptide 1 (GLP-1) receptor agonists within 12 weeks prior to visit 1 (screening)
* Anticipated change in concomitant medication known to interfere significantly with glucose metabolism, such as systemic corticosteroids, beta-blockers and MAO inhibitors
* Anticipated significant lifestyle changes during the trial according to the discretion of the trial physician, e.g. shift work (including permanent night/evening shift workers), as well as highly variable eating habits
* Cardiovascular disease, within the last 24 weeks prior to trial start, defined as: stroke; decompensated heart failure NYHA (New York Heart Association) class III or IV; myocardial infarction; unstable angina pectoris; or coronary arterial bypass graft or angioplasty
* Any clinically significant disease or disorder, except for conditions associated with type 2 diabetes, which in the trial physician's opinion could interfere with the results of the trial
* Previous participation in this trial. Participation is defined as randomised. Re-screening of screening failures is allowed only once within the limits of the recruitment period
* Known or suspected hypersensitivity to trial products or related products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 394 (Actual)
Dates: Start 2012-01-16 (Actual); Primary Completion 2012-11-19 (Actual); Study Completion 2012-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (42):
- Algeria (3):
  - Novo Nordisk Investigational Site, Algiers
  - Novo Nordisk Investigational Site, Oran
  - Novo Nordisk Investigational Site, Sétif
- Bulgaria (5):
  - Novo Nordisk Investigational Site, Haskovo
  - Novo Nordisk Investigational Site, Lukovit
  - Novo Nordisk Investigational Site, Plovdiv
  - Novo Nordisk Investigational Site, Rousse
  - Novo Nordisk Investigational Site, Sofia
- Croatia (5):
  - Novo Nordisk Investigational Site, Karlovac
  - Novo Nordisk Investigational Site, Osijek
  - Novo Nordisk Investigational Site, Rijeka
  - Novo Nordisk Investigational Site, Zadar
  - Novo Nordisk Investigational Site, Zagreb
- Czechia (3):
  - Novo Nordisk Investigational Site, Brno
  - Novo Nordisk Investigational Site, Hradec Králové
  - Novo Nordisk Investigational Site, Prague
- Germany (6):
  - Novo Nordisk Investigational Site, Bochum
  - Novo Nordisk Investigational Site, Hohenmölsen
  - Novo Nordisk Investigational Site, Rehlingen-Siersburg
  - Novo Nordisk Investigational Site, Saint Ingbert-Oberwürzbach
  - Novo Nordisk Investigational Site, Völklingen
  - Novo Nordisk Investigational Site, Wangen
- Poland (4):
  - Novo Nordisk Investigational Site, Bialystok
  - Novo Nordisk Investigational Site, Lublin
  - Novo Nordisk Investigational Site, Mazowieckie
  - Novo Nordisk Investigational Site, Warsaw
- Romania (5):
  - Novo Nordisk Investigational Site, Oradea, Bihor County
  - Novo Nordisk Investigational Site, Bucharest
  - Novo Nordisk Investigational Site, Buzău
  - Novo Nordisk Investigational Site, Galati
  - Novo Nordisk Investigational Site, Sibiu
- Slovakia (2):
  - Novo Nordisk Investigational Site, Bratislava
  - Novo Nordisk Investigational Site, Košice
- Turkey (Türkiye) (3):
  - Novo Nordisk Investigational Site, Antalya
  - Novo Nordisk Investigational Site, Istanbul
  - Novo Nordisk Investigational Site, Kocaeli
- Ukraine (6):
  - Novo Nordisk Investigational Site, Dnipro
  - Novo Nordisk Investigational Site, Kyiv
  - Novo Nordisk Investigational Site, Lviv
  - Novo Nordisk Investigational Site, Poltava
  - Novo Nordisk Investigational Site, Vinnytsia
  - Novo Nordisk Investigational Site, Zhytomyr

REFERENCES:
- [Result] Franek E, Haluzik M, Canecki Varzic S, Sargin M, Macura S, Zacho J, Christiansen JS. Twice-daily insulin degludec/insulin aspart provides superior fasting plasma glucose control and a reduced rate of hypoglycaemia compared with biphasic insulin aspart 30 in insulin-naive adults with Type 2 diabetes. Diabet Med. 2016 Apr;33(4):497-505. doi: 10.1111/dme.12982. Epub 2015 Nov 17. PMID 26435365
- [Result] Christiansen JS, Niskanen L, Rasmussen S, Johansen T, Fulcher G. Lower rates of hypoglycemia during maintenance treatment with insulin degludec/insulin aspart versus biphasic insulin aspart 30: a combined analysis of two Phase 3a studies in type 2 diabetes. J Diabetes. 2016 Sep;8(5):720-8. doi: 10.1111/1753-0407.12355. Epub 2016 Mar 6. PMID 26612062
- [Result] Haluzik M, Fulcher G, Pieber TR, Bardtrum L, Tutkunkardas D, Rodbard HW. The co-formulation of insulin degludec and insulin aspart lowers fasting plasma glucose and rates of confirmed and nocturnal hypoglycaemia, independent of baseline glycated haemoglobin levels, disease duration or body mass index: A pooled meta-analysis of phase III studies in patients with type 2 diabetes. Diabetes Obes Metab. 2018 Jul;20(7):1585-1592. doi: 10.1111/dom.13261. Epub 2018 Mar 25. PMID 29451706
- [Derived] Yang W, Akhtar S, Franek E, Haluzik M, Hirose T, Kalyanam B, Kar S, Wu T, Gogas Yavuz D, Unnikrishnan AG. Postprandial Glucose Excursions in Asian Versus Non-Asian Patients with Type 2 Diabetes: A Post Hoc Analysis of Baseline Data from Phase 3 Randomised Controlled Trials of IDegAsp. Diabetes Ther. 2022 Feb;13(2):311-323. doi: 10.1007/s13300-021-01196-7. Epub 2022 Jan 19. PMID 35044568
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 47 sites in 10 countries: Algeria (4), Bulgaria (7), Croatia (5), Czech Republic (4), Germany (5), Poland (5), Romania (5), Slovakia (3), Turkey (2), and Ukraine (7).
Pre-assignment Details: Subjects continued their metformin monotherapy or metformin in any combination with one of the following OADs: insulin secretagogue (sulphonylurea or glinide), dipeptidyl peptidase IV (DPP-IV) inhibitor, α-glucosidase inhibitors for at least 12 weeks prior to randomisation.
Groups:
- IDegAsp BID: Insulin degludec/insulin aspart (IDegAsp) was given subcutaneously twice daily (BID) with metformin. IDegAsp was given with the breakfast meal and main evening meal.
- BIAsp 30 BID: Biphasic insulin aspart 30 (BIAsp 30) was given subcutaneously twice daily (BID) with metformin. BIAsp 30 was given with the breakfast meal and main evening meal.
Period: Overall Study
Arm/Group | IDegAsp BID | BIAsp 30 BID
Started | 197 | 197
Exposed | 196 (One (1) subject was withdrawn prior to exposure due to "non fulfilment of inclusion criteria") | 195 (Two (2) subjects were withdrawn prior to exposure due to "withdrawal of consent")
Completed | 187 | 184
Not Completed | 10 | 13
Not completed — Adverse Event | 2 | 3
Not completed — Withdrawal Criteria | 3 | 0
Not completed — Unclassified | 5 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IDegAsp BID | BIAsp 30 BID | Total
Number analyzed (Participants) | 197 | 197 | 394
Age, Continuous [Mean (Standard Deviation); unit: years] — Subjects aged ≥18 years were enrolled in this study.
  years | 59.0 (9.5) | 58.8 (8.4) | 58.9 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Male and female aged ≥18 years were enrolled in this study.
  Participants
    Female | 95 | 96 | 191
    Male | 102 | 101 | 203
Glycosylated Haemoglobin (HbA1c) [Mean (Standard Deviation); unit: Percent (%) glycosylated haemoglobin] — Glycosylated haemoglobin (HbA1c) was measured at baseline.
  Percent (%) glycosylated haemoglobin | 8.5 (0.8) | 8.3 (0.7) | 8.4 (0.8)
Fasting plasma glucose (FPG) [Mean (Standard Deviation); unit: mmol/L] — Fasting plasma glucose (FPG) was measured at baseline.
  mmol/L | 10.5 (2.4) | 10.0 (2.3) | 10.2 (2.3)
Body Weight [Mean (Standard Deviation); unit: kg] — Body weight was measured at baseline.
  kg | 88.0 (15.0) | 88.5 (14.9) | 88.2 (14.9)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c (Glycosylated Haemoglobin)
Description: Change from baseline in HbA1c after 26 weeks of treatment.
Time Frame: Week 0, week 26
Population: The full analysis set (FAS) included all randomised subjects. Missing data were imputed using last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: Percent (%) glycosylated haemoglobin
Arm/Group | IDegAsp BID | BIAsp 30 BID
Number analyzed (Participants) | 197 | 197
Percent (%) glycosylated haemoglobin | -1.85 (0.97) | -1.73 (0.93)

2. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG)
Description: Change from baseline in fasting plasma glucose (FPG) after 26 weeks of treatment.
Time Frame: Week 0, week 26
Population: The full analysis set (FAS) included all randomised subjects. Missing data were imputed using LOCF. At baseline 195 subjects each in IDegAsp BID and BIAsp 30 BID treatment group were analysed.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | IDegAsp BID | BIAsp 30 BID
Number analyzed (Participants) | 195 | 195
mmol/L | -4.44 (2.97) | -3.03 (2.90)

3. Secondary Outcome: Number of Treatment Emergent Nocturnal (00:01-05:59 am) Severe or Minor Hypoglycaemic Episodes
Description: The pool of severe and minor hypoglycaemic episodes was referred to as confirmed hypoglycaemic episodes, which is presented here. Severe hypoglycaemic episodes were defined as requiring assistance to administer carbohydrate, glucagon, or other resuscitative actions. Minor hypoglycaemic episodes were defined as able to treat her/himself and plasma glucose below 3.1 mmol/L. Nocturnal hypoglycaemic episodes were defined as occurring between 00:01 and 05:59 am.
Time Frame: Onset on or after the first day of exposure to investigational product and no later than 7 days after last exposure to investigational product
Population: The safety analysis set included all subjects who received at least one dose of the investigational product or its comparator.
Measure: Number; unit: episodes
Arm/Group | IDegAsp BID | BIAsp 30 BID
Number analyzed (Participants) | 196 | 195
episodes | 60 | 260

4. Secondary Outcome: Number of Severe and Minor Treatment Emergent Hypoglycaemic Episodes
Description: The pool of severe and minor hypoglycaemic episodes was referred to as confirmed hypoglycaemic episodes, which is presented here. Severe hypoglycaemic episodes were defined as requiring assistance to administer carbohydrate, glucagon, or other resuscitative actions. Minor hypoglycaemic episodes were defined as able to treat her/himself and plasma glucose below 3.1 mmol/L.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Number; unit: episodes
Arm/Group | IDegAsp BID | BIAsp 30 BID
Number analyzed (Participants) | 196 | 195
episodes | 553 | 1221

5. Secondary Outcome: Change From Baseline in Body Weight
Description: Change from baseline in body weight after 26 weeks of treatment.
Time Frame: Week 0, week 26
Population: The safety analysis set included all subjects who received at least one dose of the investigational product or its comparator. Missing data were imputed using last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | IDegAsp BID | BIAsp 30 BID
Number analyzed (Participants) | 196 | 195
kg | 2.8 (4.1) | 2.0 (4.3)

6. Secondary Outcome: Responder for HbA1c (Below 7.0%) Without Severe and Minor Treatment Emergent Hypoglycaemic Episodes During the Last 12 Weeks of Treatment Including Only Subjects Exposed for at Least 12 Weeks
Description: Responder for HbA1c (<7.0%) without severe and minor treatment emergent hypoglycaemic episodes during the last 12 weeks of treatment. Severe + minor hypoglycaemic episodes = confirmed hypoglycaemic episodes. Severe hypoglycaemic episodes: requiring assistance to administer carbohydrate, glucagon, or other resuscitative actions. Minor hypoglycaemic episodes: able to treat her/himself and plasma glucose below 3.1 mmol/L.
Time Frame: Week 26
Population: The full analysis set (FAS) included all randomised subjects. Missing data were imputed using LOCF. Data for 15 subjects were excluded, as only subjects exposed for at least 12 weeks were included in this measurement.
Measure: Number; unit: participants
Arm/Group | IDegAsp BID | BIAsp 30 BID
Number analyzed (Participants) | 192 | 187
participants | 77 | 59

7. Secondary Outcome: Number of Treatment Emergent AEs (Adverse Events)
Description: A Treatment Emergent Adverse Event (TEAE) was defined as an event that had onset date on or after the first day of exposure to randomised treatment and no later than 7 days after the last day of randomised treatment. Severity was assessed by investigator.
Time Frame: Onset on or after the first day of exposure to investigational product and no later than 7 days after exposure to investigational product
Population: as for outcome 3
Measure: Number; unit: events
Arm/Group | IDegAsp BID | BIAsp 30 BID
Number analyzed (Participants) | 196 | 195
events
  Events | 197 | 137
  Serious | 20 | 12
  Severe | 13 | 8
  Moderate | 45 | 27
  Mild | 139 | 102
  Fatal | 2 | 2

ADVERSE EVENTS:
Time Frame: From the first trial-related activity after the subject had signed the informed consent (Week -1) and until post-treatment follow-up period (Week 27).
Description: The safety analysis set included all subjects who received at least one dose of the investigational product or its comparator.
Arm/Group | IDegAsp BID | BIAsp 30 BID
Serious Adverse Events (participants affected / at risk) | 13/196 | 10/195
Other Adverse Events (participants affected / at risk) | 15/196 | 7/195
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDegAsp BID (N=196) | BIAsp 30 BID (N=195)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery insufficiency (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 2 (2)
Deafness neurosensory (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Optic ischaemic neuropathy (Eye disorders) | 0 (0) | 1 (1)
Colonic stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia, obstructive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Meningitis pneumococcal (Infections and infestations) | 1 (1) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Colon cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Hypoglycaemic unconsciousness (Nervous system disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDegAsp BID (N=196) | BIAsp 30 BID (N=195)
Nasopharyngitis (Infections and infestations) | 15 (17) | 7 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk maintains the right to be informed of any Investigator plans for publication and to review any scientific paper, presentation, communication or other information concerning the investigation described in this protocol. Any such communication must be submitted in writing to the Novo Nordisk trial manager prior to submission for comments. Comments will be given within four weeks from receipt of the planned communication.